CLINICAL TRIAL: NCT04549168
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 3 Study of the Efficacy and Safety of Lemborexant in Chinese Subjects With Insomnia Disorder
Brief Title: A Study of Lemborexant in Chinese Participants With Insomnia Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2006-J086-311
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2023-05

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Insomnia disorder; Lemborexant; Chinese Participants; E2006
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — lemborexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lemborexant 10 mg (Experimental): Participants will receive one lemborexant 10 mg tablet, orally, once daily for 30 consecutive nights on each night approximately 5 minutes before participants intends to try to sleep.
  Interventions: Drug: Lemborexant
- Placebo (Placebo Comparator): Participants will receive one placebo matched to lemborexant 10 mg tablet, orally, once daily for 30 consecutive nights on each night approximately 5 minutes before participants intends to try to sleep.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lemborexant — Lemborexant 10 mg tablet.
  Other Names: E2006
  Arms: Lemborexant 10 mg
Drug: Placebo — Placebo tablet matched to lemborexant 10 mg tablet.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to confirm using polysomnography (PSG) that lemborexant 10 milligram (mg) is superior to placebo on objective sleep onset as assessed by latency to persistent sleep (LPS) during the last 2 nights of 1 month of treatment in participants with insomnia disorder.

DETAILED DESCRIPTION:
The study will have 2 phases: the Prerandomization Phase and the Randomization Phase. The Prerandomization Phase will comprise 3 periods that will last up to a maximum of 35 days: a Screening Period, a Run-in Period, and a Baseline Period. The Randomization Phase will comprise a Treatment Period during which participants will be treated for 30 nights (1 month) and a minimum 14-day Follow-up Period before an End of Study (EOS) Visit (up to 54 days). The total study duration for each participant on this study is 89 days.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in this study:

1. Chinese male or female, age 18 years or older, at the time of informed consent (in Taiwan only participants with age 20 years or older are eligible)
2. Meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for Insomnia Disorder, as follows:

   * Complains of dissatisfaction with night time sleep, in the form of difficulty staying asleep and/or awakening earlier in the morning than desired despite adequate opportunity for sleep
   * Frequency of complaint greater than or equal to (>=) 3 times per week
   * Duration of complaint >=3 months
   * Associated with complaint of daytime impairment
3. At Screening: History of sSOL >=30 minutes on at least 3 nights per week in the previous 4 weeks and/or sWASO >=60 minutes on at least 3 nights per week in the previous 4 weeks
4. At Screening: Reports regular time spent in bed, either sleeping or trying to sleep, between 7 and 9 hours
5. At second Screening Visit (Visit 2a) and Run-in Visit (Visit 3a): Sleep diary confirms regular bedtime, defined as the time the participant attempts to sleep, between 21:00 and 01:00 on at least 5 of the final 7 nights and regular waketime, defined as the time the participant gets out of bed for the day, between 05:00 and 10:00 on at least 5 of the final 7 nights
6. At Screening and Baseline: ISI score >=15
7. Confirmation of current insomnia symptoms, as determined from responses on the sleep diary on the 7 most recent mornings before the first PSG during Screening Period (Visit 2a) and Run-in visit (Visit 3a), such that sSOL >=30 minutes on at least 3 of the 7 nights and/or sWASO >=60 minutes on at least 3 of the 7 nights
8. At the second Screening Visit (Visit 2a) and the Run-in visit (Visit 3a): Confirmation of sufficient duration of time spent in bed, as determined from responses on the sleep diary on the 7 most recent mornings before the Visit, such that there are no more than 2 nights with time spent in bed duration less than (<) 7 hours or greater than (>) 10 hours
9. During the Run-in Period, objective (PSG) evidence of insomnia as follows:

   1. LPS average >=30 minutes on the 2 consecutive Baseline PSGs, with neither night <20 minutes and/or
   2. WASO average >=60 minutes on the two consecutive Baseline PSGs, with neither night <45 minutes
10. Willing and able to comply with all aspects of the protocol, including staying in bed for at least 7 hours each night
11. Willing not to start a behavioral or other treatment program for the treatment of insomnia during the participant's participation in the study

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from this study:

1. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin test). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug
2. Females of childbearing potential who: Within 28 days before study entry, did not use a highly effective method of contraception, which includes any of the following:

   * total abstinence (if it is their preferred and usual lifestyle)
   * an intrauterine device or intrauterine hormone-releasing system
   * a contraceptive implant
   * an oral contraceptive (participant must be on a stable dose of the same oral contraceptive product for at least 28 days before dosing and throughout the study and for 28 days after study drug discontinuation)
   * have a vasectomized partner with confirmed azoospermia
   * do not agree to use a highly effective method of contraception (as described above) throughout the entire study period and for 28 days after study drug discontinuation It is permissible that if a highly effective method of contraception is not appropriate or acceptable to the participant, then the participant must agree to use a medically acceptable method of contraception, that is, double-barrier methods of contraception such as latex or synthetic condom plus diaphragm or cervical/vault cap with spermicide NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (that is, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing)
3. Any history of a medical or psychiatric condition that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
4. A prolonged corrected QT interval by Fredericia's formula (QTcF) interval (QTcF >450 millisecond [ms]) as demonstrated by a repeated electrocardiogram. A history of risk factors for torsade de pointes (for example, heart failure, hypokalemia, family history of long QT Syndrome) or the use of concomitant medications that prolonged the QTcF interval
5. Any suicidal ideation with intent with or without a plan at Screening or within 6 months of Screening
6. Any suicidal behavior in the past 10 years
7. Evidence of clinically significant disease (for example, cardiac; respiratory including chronic obstructive pulmonary disease, acute and/or severe respiratory depression; gastrointestinal; moderate and severe hepatic impairment; renal including severe renal impairment; neurological including myasthenia gravis; psychiatric disease; or malignancy within the past 5 years other than adequately treated basal cell carcinoma) or chronic pain that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments. Participants for whom a sedating drug would be contraindicated for safety reasons because of the participant's occupation or activities are also excluded
8. Hypersensitivity to lemborexant or to their excipients
9. Scheduled for surgery during the study
10. Known to be human immunodeficiency virus positive
11. Active viral hepatitis (B or C) as demonstrated by positive serology
12. History of drug or alcohol dependency or abuse within approximately the last 2 years
13. A current diagnosis of sleep-related breathing disorder including obstructive sleep apnea (with or without continuous positive airway pressure treatment), periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep disorder, or narcolepsy, or an exclusionary score on screening instruments to rule out individuals with symptoms of certain sleep disorders other than insomnia as follows:

    * Snoring, Tiredness, Observed apnea, high blood Pressure (STOP)-Body mass index (BMI), Age, Neck circumference, and Gender (BANG) score >=5
    * International Restless Legs Scale score >=16
14. Apnea-hypopnea Index >15 or Periodic Limb Movement with Arousal Index >15 as measured on the PSG at the second Screening Visit
15. Reports symptoms potentially related to narcolepsy, that in the clinical opinion of the investigator indicates the need for referral for a diagnostic evaluation for the presence of narcolepsy
16. Reports a history of sleep-related violent behavior, or sleep driving, or any other complex sleep-related behavior (for example, making phone calls or preparing and eating food while sleeping)
17. For participants who underwent diagnostic PSG within 1 year before informed consent:

    * Age 18 to 64 years: Apnea Hypopnea Index >=10, or Periodic Limb Movements with Arousal Index >=10
    * Age >=65 years: Apnea Hypopnea Index >15, or Periodic Limb Movements with Arousal Index >15
18. Beck Depression Inventory-II score >19 at Screening
19. Beck Anxiety Inventory score >15 at Screening
20. Habitually naps during the day more than 3 times per week
21. Excessive caffeine use that in the opinion of the investigator contributes to the participant's insomnia, or habitually consumes caffeine containing beverages after 18:00 and is unwilling to forego caffeine after 18:00 for the duration of his/her participation in the study. Participants are excluded if, in the previous 3 months, they had symptoms that would meet DSM-5 criteria for caffeine intoxication, which includes consumption of a high dose of caffeine (significantly in excess of 250 mg) and >=5 of the following symptoms: restlessness, nervousness, excitement, insomnia, flushed face, diuresis, gastrointestinal disturbance, muscle twitching, rambling flow of thought and speech, tachycardia or cardiac arrhythmia, periods of high energy, or psychomotor agitation. To be exclusionary, those symptoms must cause distress or impairment in social, occupational and other forms of functioning, and not be associated with other substance, mental disorder or medical condition
22. Reports habitually consuming more than 14 drinks containing alcohol per week (females) or more than 21 drinks containing alcohol per week (males), or unwilling to limit alcohol intake to no more than 2 drinks per day or forego having alcohol within the 3 hours before bedtime for the duration of his/her participation in the study
23. Excluding comorbid nocturia that is causing or exacerbating the insomnia
24. Used any prohibited prescription or over-the-counter concomitant medications within 1 week or 5 half-lives, whichever is longer, before the first dose of study medication (Run-in Period)
25. Used any modality of treatment for insomnia, including cognitive behavioral therapy or marijuana within 1 week or 5 half-lives, whichever is longer, before the first dose of study medication (Run-in Period)
26. Failed treatment with dual orexin receptor antagonist drugs (efficacy and/or safety) following treatment with an appropriate dose and of adequate duration in the opinion of the investigator
27. Transmeridian travel across more than 3 time zones in the 2 weeks before Screening, or between Screening and Baseline, or plans to travel across more than 3 time zones during the study (China mainland will be considered as 1 time zone)
28. A positive drug test at Screening, Run-in, or Baseline, or unwilling to refrain from use of recreational drugs during the study
29. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days or 5 half-lives, whichever is longer preceding informed consent
30. Previously participated in any clinical trial of lemborexant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- China (21):
  - Beijing Tiantan Hosptial, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Mental Health Center, Xinxiang, Henan
  - Wuhan Mental Health Center, Wuhan, Hubei
  - Nanjing Brain Hosptial, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin First University Affiliated Hospital, Changchun, Jilin
  - Inner Mongolia Autonomous Region Peoples Hospital, Hohhot, Mongolia
  - Tangdu Hospital, Xi'an, Shaanxi
  - Shandong Provincial Qianfushan Hospital, Jinan, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shannxi
  - Tianjin Anding Hospital, Tianjin, Tianjin Municipality
- Taiwan (2):
  - Chang Gung Medical Foundation Linkou Chang Gung Memorial Hospital, Taoyuan, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Mi WF, Wen D, Xu L, Pan J, Gu P, Wang C, Tang J, Zhang L, Liu CF, Yuan C, Wang H, Yamakawa N, Takase T, Moline M, Lu L. A phase 3, multicenter, double-blind, randomized, placebo-controlled clinical trial of lemborexant in adults with insomnia disorder. Sleep Med. 2025 Dec 18;139:108722. doi: 10.1016/j.sleep.2025.108722. Online ahead of print. PMID 41442783

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 21 sites in China mainland and 2 sites in Taiwan from 06 November 2020 to 17 March 2023.
Pre-assignment Details: The study consisted of two phases: the prerandomization phase and the randomization phase. A total of 194 participants were enrolled in pre-randomization phase and then went on to randomization phase to receive study treatment.
Groups:
- Prerandomization Phase: All Participants: Participants received one lemborexant-matched placebo tablet, orally, once daily 5 minutes before bedtime at Day -10 until Day -2.
- Randomization Phase: Placebo: Participants received one lemborexant-matched placebo tablet, orally, once daily 5 minutes before bedtime at Day 1 until Day 31 (or for 30 consecutive nights) during the Treatment Period and were followed up to Day 44.
- Randomization Phase: Lemborexant 10 mg: Participants received one lemborexant 10 milligrams (mg) tablet, orally, once daily 5 minutes before bedtime at Day 1 until Day 31 (or for 30 consecutive nights) during the Treatment Period and were followed up to Day 44.
Period: Prerandomization Phase
Arm/Group | Prerandomization Phase: All Participants | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Started | 194 | 0 | 0
Completed | 194 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Randomization Phase
Arm/Group | Prerandomization Phase: All Participants | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Started | 0 | 100 | 94
Full Analysis Set (FAS) (The FAS was the group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose primary efficacy measurement.) | 0 | 100 | 93
Completed | 0 | 96 | 92
Not Completed | 0 | 4 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Other | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set was the group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose safety assessment.
Groups:
- Randomization Phase: Lemborexant 10 mg: Participants received one lemborexant 10 mg tablet, orally, once daily 5 minutes before bedtime at Day 1 until Day 31 (or for 30 consecutive nights) during the Treatment Period and were followed up to Day 44.
- Total: Total of all reporting groups
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg | Total
Number analyzed (Participants) | 100 | 94 | 194
Age, Customized [Count of Participants; unit: Participants]
  <55 years old | 78 | 73 | 151
  >=55 - <65 years old | 14 | 19 | 33
  >=65 - <75 years old | 8 | 2 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 58 | 132
  Male | 26 | 36 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 100 | 94 | 194
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 100 | 94 | 194

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Mean Latency to Persistent Sleep (LPS) Over the Last 2 Nights of 1 Month of Treatment of Lemborexant 10 mg Compared to Placebo
Description: LPS was defined as the time in minutes from lights off to the first epoch of 20 consecutive epochs of non- wakefulness as measured by polysomnography (PSG). Change from baseline to average LPS on Days 29 and 30 was reported. The outcome measure was planned to be assessed for randomization phase only.
Time Frame: Baseline, Days 29 and 30
Population: The FAS was the group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose primary efficacy measurement. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Number analyzed (Participants) | 89 | 84
minutes | -21.71 (42.809) | -39.47 (46.147)
Statistical Analysis 1: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.0585, MMRM — Data was analyzed using mixed effect model repeated measurement analysis (MMRM), and the missing values were imputed using multiple imputation and assumed to be missing not at random (MNAR); LS geometric mean ratio = 0.795, 95% CI 2-sided [0.627 to 1.008]

2. Secondary Outcome: Change From Baseline of Mean Objective Sleep Efficiency (SE) Over the Last 2 Nights of 1 Month Treatment of Lemborexant 10 mg Compared to Placebo
Description: SE was defined as percentage (%) of time spent in bed asleep, calculated as total sleep time (TST) divided by interval from lights off until lights on as measured by PSG multiplied by 100. Change from baseline to average SE on Days 29 and 30 was reported. The outcome measure was planned to be assessed for randomization phase only.
Time Frame: Baseline, Days 29 and 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % time (minutes) in bed asleep
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Number analyzed (Participants) | 89 | 84
% time (minutes) in bed asleep | 7.40 (12.853) | 15.33 (11.124)
Statistical Analysis 1: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — Data was analyzed using MMRM, and the missing values were imputed using multiple imputation and assumed to be MNAR; LSM difference = 7.10, 95% CI 2-sided [4.39 to 9.81]

3. Secondary Outcome: Change From Baseline in Mean Objective Wake After Sleep Onset (WASO) Over the Last 2 Nights of 1 Month Treatment of Lemborexant 10 mg Compared to Placebo
Description: WASO was defined as minutes of wake from the onset of persistent sleep until lights on as measured by PSG. Change from baseline to average WASO on Days 29 and 30 was reported. The outcome measure was planned to be assessed for randomization phase only.
Time Frame: Baseline, Days 29 and 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Number analyzed (Participants) | 89 | 84
minutes | -14.30 (42.733) | -36.65 (35.342)
Statistical Analysis 1: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.0002, MMRM — Data was analyzed using MMRM, and the missing values were imputed using multiple imputation and assumed to be MNAR; LSM difference = -17.84, 95% CI 2-sided [-27.16 to -8.51]

4. Secondary Outcome: Change From Baseline of Subjective Sleep Onset Latency (sSOL) Over the Last 7 Nights of 1 Month Treatment of Lemborexant 10 mg Compared to Placebo
Description: sSOL was defined as estimated minutes from the time that the participant attempted to sleep until sleep onset. Change from baseline to average sSOL of Nights 24 to 30 was reported. The outcome measure was planned to be assessed for randomization phase only.
Time Frame: Baseline, Nights 24 to 30
Population: The FAS was the group of randomized participants who received at least one dose of randomized study drug and had at least one postdose primary efficacy measurement. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Number analyzed (Participants) | 98 | 91
minutes | -22.41 (32.183) | -33.10 (50.060)
Statistical Analysis 1: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.0063, MMRM — Data was analyzed using MMRM, and the missing values were imputed using multiple imputation and assumed to be MNAR; LS geometric mean ratio = 0.776, 95% CI 2-sided [0.647 to 0.930]

5. Secondary Outcome: Change From Baseline of Subjective Sleep Efficiency (sSE) Over the Last 7 Nights of 1 Month of Treatment of Lemborexant 10 mg Compared to Placebo
Description: sSE was defined as percentage of subjective total sleep time (sTST) divided by subjective time spent in bed, calculated as the interval from the time the participant reported attempting to sleep until the time participant stopped trying to sleep for the night (operationalized as the time the participant got out of bed for the day), and time spent asleep derived from subjective time spent in bed minus subjective wake after sleep onset (sWASO). WASO: estimated minutes of wake at night after initial sleep onset to time stopped trying to sleep for the night. Change from baseline to average sSE of Nights 24 to 30 was reported. The outcome measure was planned to be assessed for randomization phase only.
Time Frame: Baseline, Nights 24 to 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % of time (minutes) in bed asleep
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Number analyzed (Participants) | 95 | 84
% of time (minutes) in bed asleep | 8.88 (11.630) | 13.16 (16.559)
Statistical Analysis 1: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.0242, MMRM — Data was analyzed using MMRM, and the missing values were imputed using multiple imputation and assumed to be MNAR; LSM difference = 4.49, 95% CI 2-sided [0.59 to 8.39]

6. Secondary Outcome: Change From Baseline in Subjective Wake After Sleep Onset Over the Last 7 Nights of 1 Month Treatment of Lemborexant 10 mg Compared to Placebo
Description: sWASO was defined as sum of estimated minutes of wake during the night after initial sleep onset until the time the participant stopped trying to sleep for the night, operationalized as the time the participant got out of bed for the day. Change from baseline to average sWASO of Nights 24 to 30 was reported. The outcome measure was planned to be assessed for randomization phase only.
Time Frame: Baseline, Nights 24 to 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Number analyzed (Participants) | 97 | 88
minutes | -22.39 (48.620) | -32.14 (60.110)
Statistical Analysis 1: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.1625, MMRM — Data was analyzed using MMRM, and the missing values were imputed using multiple imputation and assumed to be MNAR; LSM difference = -10.36, 95% CI 2-sided [-24.95 to 4.22]

7. Secondary Outcome: Change From Baseline of Mean Latency to Persistent Sleep Over the First 2 Nights of 1 Month of Treatment of Lemborexant 10 mg Compared to Placebo
Description: LPS was defined as the time in minutes from lights off to the first epoch of 20 consecutive epochs of non- wakefulness as measured by polysomnography. Change from baseline to average LPS on Nights 1 and 2 was reported. The outcome measure was planned to be assessed for randomization phase only.
Time Frame: Baseline, Nights 1 and 2
Population: The FAS was the group of randomized participants who received at least one dose of randomized study drug and had at least one postdose primary efficacy measurement.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Number analyzed (Participants) | 100 | 93
minutes | -16.52 (42.970) | -34.64 (48.102)
Statistical Analysis 1: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.0515, MMRM — Data was analyzed using MMRM, and the missing values were imputed using multiple imputation and assumed to be MNAR; LS geometric mean ratio = 0.815, 95% CI 2-sided [0.663 to 1.001]

8. Secondary Outcome: Change From Baseline of Mean Sleep Efficiency Over the First 2 Nights of 1 Month of Treatment of Lemborexant 10 mg Compared to Placebo
Description: SE was defined as percentage of time spent in bed asleep, calculated as total sleep time divided by interval from lights off until lights on as measured by PSG, multiplied by 100. Change from baseline to average SE on Nights 1 and 2 was reported. The outcome measure was planned to be assessed for randomization phase only.
Time Frame: Baseline, Nights 1 and 2
Population: The FAS was the group of randomized participants who received at least 1 dose of randomized study drug and had at least 1 postdose primary efficacy measurement.
Measure: Mean (Standard Deviation); unit: % of time (minutes) in bed asleep
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Number analyzed (Participants) | 100 | 93
% of time (minutes) in bed asleep | 6.99 (9.595) | 15.58 (11.725)
Statistical Analysis 1: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — Data was analyzed using MMRM, and the missing values were imputed using multiple imputation and assumed to be MNAR; LSM difference = 7.74, 95% CI 2-sided [5.61 to 9.86]

9. Secondary Outcome: Change From Baseline of Mean Wake After Sleep Onset Over the First 2 Nights of 1 Month of Treatment of Lemborexant 10 mg Compared to Placebo
Description: WASO was defined as minutes of wake from the onset of persistent sleep until lights on as measured by PSG. Change from baseline to average WASO on Nights 1 and 2 was reported. The outcome measure was planned to be assessed for randomization phase only.
Time Frame: Baseline, Nights 1 and 2
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Number analyzed (Participants) | 100 | 93
minutes | -17.99 (29.782) | -42.86 (35.970)
Statistical Analysis 1: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p < 0.0001, MMRM — Data was analyzed using MMRM, and the missing values were imputed using multiple imputation and assumed to be MNAR; LSM difference = -21.25, 95% CI 2-sided [-28.15 to -14.35]

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE was defined as an AE with onset date on or after the first dose of study drug up to 14 days after the last dose of study drug. An SAE was any untoward medical occurrence that at any dose: resulted in death, was life-threatening (that is, participant was at immediate risk of death from AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug). The outcome measure was planned to be assessed for randomization phase only.
Time Frame: From the first dose of study drug up to 44 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Number analyzed (Participants) | 100 | 94
Participants
  TEAEs | 21 | 30
  Serious TEAEs | 1 | 0

11. Secondary Outcome: Change From Baseline in Insomnia Severity Index (ISI) Total Score After 1 Month of Treatment With Lemborexant 10 mg Compared to Placebo
Description: The ISI was a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia. The 7 dimensions evaluated are severity of: sleep onset; sleep maintenance; early-morning awakening problems; sleep dissatisfaction; interference of sleep difficulties with daytime functioning; noticeability of the sleep problems by others; and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (from 0= no problem, 1= satisfied, 2= moderately satisfied, 3= dissatisfied and 4=very severe problem). Total ISI score was calculated as sum of scores of all 7 individual items, ranging between 0 to 28. A higher score indicated more severe illness. The outcome measure was planned to be assessed for randomization phase only.
Time Frame: Baseline to Day 31
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Number analyzed (Participants) | 89 | 87
Score on a scale | -6.48 (5.246) | -9.64 (5.528)
Statistical Analysis 1: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.0006, ANCOVA — Based on Analysis of Covariance (ANCOVA) model with factors of age group, site, treatment, and the baseline ISI as a covariate; LSM difference = -2.85, 95% CI 2-sided [-4.45 to -1.25], Standard Error of Mean 0.811

12. Secondary Outcome: Change From Baseline in Insomnia Severity Index Daytime Functioning Score After 1 Month of Treatment With Lemborexant 10 mg Compared to Placebo
Description: The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia. The 4 dimensions out of 7 evaluated for daily functioning are severity of: sleep dissatisfaction; interference of sleep difficulties with daytime functioning; noticeability of the sleep problems by others; and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (from 0= no problem, 1= satisfied, 2= moderately satisfied, 3= dissatisfied and 4=very severe problem), Daytime Functioning score was calculated as sum of scores of item 4 to 7, ranging between 0 to 16. A higher score indicated more severe illness. The outcome measure was planned to be assessed for randomization phase only.
Time Frame: Baseline to Day 31
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Number analyzed (Participants) | 89 | 87
Score on a scale | -3.76 (3.093) | -5.77 (3.510)
Statistical Analysis 1: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.0005, ANCOVA — Based on ANCOVA model with factors of age group, site, treatment, and the baseline ISI as a covariate; LSM difference = -1.74, 95% CI 2-sided [-2.70 to -0.78], Standard Error of Mean 0.488

13. Secondary Outcome: Number of Participants With Rebound Insomnia on Average of First 3 Nights (Nights 31 to 33), Average of First 7 Nights (Nights 31 to 37), and Average of Last 7 Nights (Nights 38 to 44) During the Follow-up Period
Description: Rebound insomnia was defined as worsened sleep relative to screening after study drug treatment was completed. Sleep diary data from the follow-up period was compared to sleep diary data from the screening period to assess whether participants experience rebound insomnia. Number of participants with rebound insomnia assessed by sleep diary (sSOL and sWASO) was reported. The outcome measure was planned to be assessed for randomization phase only.
Time Frame: First 3 nights (Nights 31 to 33), First 7 nights (Nights 31 to 37) and Last 7 nights (Nights 38 to 44) of Follow up Period
Population: The FAS was the group of randomized participants who received at least one dose of randomized study drug and had at least one postdose primary efficacy measurement. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. Here "number analyzed" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Number analyzed (Participants) | 94 | 91
Participants
  sSOL, Average of First 3 nights of follow-up period | 5 | 7
  sSOL, Average of First 7 nights of follow-up period | 6 | 7
  sSOL, Average of Last 7 nights of follow-up period: number analyzed (Participants) | 94 | 89
  sSOL, Average of Last 7 nights of follow-up period | 9 | 11
  sWASO, Average of First 3 nights of follow-up period | 15 | 10
  sWASO, Average First 7 nights of follow-up period | 13 | 12
  sWASO, Average of Last 7 nights of follow-up period: number analyzed (Participants) | 94 | 89
  sWASO, Average of Last 7 nights of follow-up period | 8 | 12

14. Secondary Outcome: Change From Baseline in Mean Morning Residual Sleepiness Score Evaluated During Treatment and Follow-up Periods
Description: The Sleep Diary was used to assess subjective ratings of morning sleepiness with the following question: "How sleepy/alert do you feel this morning?" Participants rated their sleepiness/alertness level on a Likert scale from 1 to 9, with 1 being extremely poor (sleepy) and 9 being extremely good (alert). Higher score indicated better outcome. Change from baseline of the morning sleepiness item on the sleep diary for the average of first 7 mornings and the average of last 7 mornings of the Treatment Period; and the average of the first 7 mornings and the average of the last 7 mornings of the Follow-up Period was reported. The outcome measure was planned to be assessed for randomization phase only.
Time Frame: Baseline, First 7 mornings (Mornings 1 to 7) and Last 7 mornings (Mornings 24 to 30) of Treatment period; First 7 mornings (Mornings 31 to 37) and Last 7 mornings (Mornings 38 to 44) of Follow-up period
Population: The FAS was the group of randomized participants who received at least one dose of randomized study drug and had at least one postdose primary efficacy measurement. Here "number analyzed" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
Number analyzed (Participants) | 100 | 93
Score on a scale
  First 7 mornings of treatment period | 0.20 (0.982) | 0.59 (1.284)
  Last 7 mornings of treatment period: number analyzed (Participants) | 98 | 91
  Last 7 mornings of treatment period | 0.75 (1.577) | 1.15 (1.625)
  First 7 mornings of follow-up period: number analyzed (Participants) | 94 | 90
  First 7 mornings of follow-up period | 0.81 (1.508) | 1.18 (1.534)
  Last 7 mornings of follow-up period: number analyzed (Participants) | 93 | 89
  Last 7 mornings of follow-up period | 0.91 (1.682) | 1.22 (1.434)
Statistical Analysis 1: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.0312, MMRM — Data was analyzed using MMRM, and the missing values were imputed using multiple imputation and assumed to be MNAR; LSM difference = 0.34, 95% CI 2-sided [0.03 to 0.65] — First 7 mornings of treatment period
Statistical Analysis 2: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.1460, MMRM — Data was analyzed using MMRM, and the missing values were imputed using multiple imputation and assumed to be MNAR; LSM difference = 0.32, 95% CI 2-sided [-0.11 to 0.76] — Last 7 mornings of treatment period
Statistical Analysis 3: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.1613, MMRM — Data was analyzed using MMRM, and the missing values were imputed using multiple imputation and assumed to be MNAR; LSM difference = 0.29, 95% CI 2-sided [-0.12 to 0.70] — First 7 mornings of follow-up period
Statistical Analysis 4: Comparison: Randomization Phase: Placebo vs Randomization Phase: Lemborexant 10 mg; Test type: Superiority; p = 0.2852, MMRM — Data was analyzed using MMRM, and the missing values were imputed using multiple imputation and assumed to be MNAR; LSM difference = 0.23, 95% CI 2-sided [-0.19 to 0.65] — Last 7 mornings of follow-up period

ADVERSE EVENTS:
Time Frame: From signing of the consent form up to 79 days which include 35 days for prerandomization phase and up to 44 days for randomization phase
Description: Adverse events were reported for prerandomization and randomization phase.
Arm/Group | Prerandomization Phase: All Participants | Randomization Phase: Placebo | Randomization Phase: Lemborexant 10 mg
All-Cause Mortality (participants affected / at risk) | 0/194 | 0/100 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/194 | 1/100 | 0/94
Other Adverse Events (participants affected / at risk) | 19/194 | 20/100 | 30/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Prerandomization Phase: All Participants (N=194) | Randomization Phase: Placebo (N=100) | Randomization Phase: Lemborexant 10 mg (N=94)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prerandomization Phase: All Participants (N=194) | Randomization Phase: Placebo (N=100) | Randomization Phase: Lemborexant 10 mg (N=94)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 3 | 3 | 8
Influenza (Infections and infestations) | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 1
Blood cholesterol increased (Investigations) | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Electrocardiogram ST-T segment abnormal (Investigations) | 1 | 1 | 0
Haemoglobin urine present (Investigations) | 0 | 1 | 0
Red blood cells urine positive (Investigations) | 0 | 1 | 0
Urine ketone body present (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1
Sleep paralysis (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT04549168/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT04549168/SAP_001.pdf